CLINICAL TRIAL: NCT06892236
Title: Preparation of Large-scale Patient-specific Induced Pluripotent Stem Cells (iPSC) Library for Cell Gene Editing for the Treatment of Alpha1-antitrypsin Deficiency
Brief Title: Preparation of IPSC for Cell Gene Editing for the Treatment of AATD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Stefania Ottaviani, Researcher, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AATD-iPSC
Record Dates: First submitted 2025-02-24; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- severe AATD patients (Other): blood samples from severe AATD patients to obtain iPSC cells
  Interventions: Genetic: iPSC generation

INTERVENTIONS:
Genetic: iPSC generation — Base editing

SUMMARY:
Alpha 1-antitrypsin (AAT) deficiency is a genetic condition that leads to lung and/or liver diseases; current treatment of weekly augmentation of AAT addresses only lung diseases with moderate efficacy. Novel treatments based on gene editing can restore physiological levels of AAT and address lung and liver disease.

The aim is to generate induced pluripotent stem cells (iPSC) from blood and urine of patients with different severe Alpha1-antitrypsin deficiency (AATD) genotypes. Further, the iPSC will be differentiated into hepatocytes (iHep). Since hepatocytes are the main producers of AAT, the iHep will be used to test different approaches of gene editing to correct various mutations. Gene editing will be conducted at University of Bern (Switzerland)

DETAILED DESCRIPTION:
AAT is majorly produced in the hepatocytes therefore correction in the hepatocyte is a most promising approach. iHep cells as well as pluripotent stem cell or mesenchymal stem cell-derived hepatocyte-like cells provide potential cell sources for disease modeling, transplantation, and tissue engineering independent of donor organs.

However, all the studies reported in the literature, including the large drug library screening, are based on one or few AAT variant or at most few hiPSC cell lines derived from AATD patients. Moreover, only a subgroup of 10% of PI*ZZ developed a clinically relevant liver disease and there is a strong suspect that genetic and/or environmental modifiers determine whether an affected homozygote is susceptible to liver disease. Moreover, there is no study about the efficacy of potential drug in reducing cellular AAT accumulation for other AAT genotypes rather than PI*ZZ and for other rare mutations associated with liver inclusions and clinically apparent liver disease. This limitation represents a strong barrier in the development of new therapies. For this reason, the investigators will select candidates with different disease profiles. The investigators plan to recruit patients with different genotypes, including the carriers of rare pathological variants. iPSC will be generated from peripheral blood and urine cells, then cells will be characterised and stored. The PBMC will be frozen and will be reprogrammed to Induced pluripotent stem cells. The derived IPSC will be characterized by standard methods of immunofluroscence, qRTPCR, combined genomic hybridization (CGH) and flowcytometry, and will be differentiated to three germ layers.

Further, the investigators will differentiate iPSC into hepathocytes (iHep). The iPSC derived hepatocytes from the AAT deficient patients will be characterized for the mutations. There have been attempts to develop hepatocyte specific targeting but with limitations therefore in the current proposal the investigators aim at developing and testing two different approaches for cell specific targeting: 1) by hepatocyte specific liposome/virosome by integrating/conjugating asialofeutin on the surface of the liposome/virosomes either as protein fragments or peptides; 2) coating the liposome/virosome carrying the BEs with hepatocyte derived exovesicle surface membrane and delivering the BEs in the AATD iHep to test the feasibility of this method for treatment of AAT deficiency. These hepatocytes will be treated with BEs and its effect will be evaluated by deep sequencing, immunohistochemistry and secretion of AAT will be confirmed by ELISA.

Base editing is an emerging method of precision medicine that the investigators are going to use as treatment to cure AATD. In order to reach the target, the investigators propose here to use extracellular vesicles to deliver base editors in the liver. Extracellular vesicles are secreted by almost all types of cells and can be used as carriers of potential therapeutic proteins. It has been shown that base editing is a very promising technique to correct genetic mutation. However, several challenges remain unresolved and, in this grant, the investigators want to address: specificity, stability, bio-distribution, and analysis of long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years at the time of signing the ICF
* diagnosis of severe AATD (2 pathological variants)

Exclusion Criteria:

* incapability to give informed consent
* subject under augmentation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of severe AATD patients included in the study | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Sc Pneumologia, Pavia, Pavia, Italy